CLINICAL TRIAL: NCT01344187
Title: A Multi-Center, Randomized, Placebo-Controlled Evaluation of the Safety and Efficacy of the KXL System With VibeX (Riboflavin Ophthalmic Solution) for Corneal Collagen Cross-Linking in Eyes With Keratoconus
Brief Title: Safety and Efficacy Study of Corneal Collagen Cross-Linking in Eyes With Keratoconus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KXL-001
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- riboflavin solution and KXL System (Experimental): Subjects will receive riboflavin solution followed by UVA irradiation for 4 minutes
  Interventions: Drug: riboflavin solution; Device: KXL System
- placebo solution and KXL System (Placebo Comparator): Subjects will receive placebo solution followed by UVA irradiation for 4 minutes
  Interventions: Drug: placebo solution; Device: KXL System

INTERVENTIONS:
Drug: riboflavin solution — 0.12% riboflavin ophthalmic solution
  Other Names: VibeX
  Arms: riboflavin solution and KXL System
Drug: placebo solution — 0.0% riboflavin ophthalmic solution
  Other Names: placebo
  Arms: placebo solution and KXL System
Device: KXL System — 30 mW/cm2
  Other Names: UVA Irradiation

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of corneal collagen cross-linking performed with VibeX (riboflavin ophthalmic solution) and the KXL System as compared to placebo in impeding the progression of, and/or reducing, maximum corneal curvature.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria in order to be enrolled into the trial:

1. Be at least 12 years of age, male or female, of any race;
2. Provide written informed consent and sign a HIPAA form. Patients who are under the age of 18 will need to sign an assent form as well as having a parent or legal guardian sign an informed consent;
3. Willingness and ability to follow all instructions and comply with schedule for follow-up visits;
4. For females capable of becoming pregnant, agree to have urine pregnancy testing performed prior to randomization of the study eye and prior to treatment of a fellow and/or cross-over eye; must not be lactating, and must agree to use a medically acceptable form of birth control for at least one week prior to the randomization visit, one week prior to treatment of a fellow eye or cross-over eye, and continue to use the method for one month following the last treatment. Acceptable forms for birth control are spermicide with barrier, oral contraceptive, injectable or implantable method of contraception, transdermal contraceptive, intrauterine device, or surgical sterilization of partner. For non-sexually active females, abstinence will be considered an acceptable form of birth control. Women considered capable of becoming pregnant include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (e.g. hysterectomy, bilateral tubal ligation, or bilateral oophorectomy);
5. Having topographic evidence of keratoconus with a diagnosis of mild, moderate, or severe keratoconus defined as the following:

   * Mild Keratoconus:

     * Axial topography consistent with keratoconus
     * Flat Pentacam keratometry reading ≤ 51.00D
   * Moderate Keratoconus:

     * Axial topography consistent with keratoconus
     * Flat Pentacam keratometry reading ≥ 51.01 D and ≤ 56.00 D or astigmatism ≥ 8.00 D
   * Severe Keratoconus:

     * Axial topography consistent with keratoconus with marked areas of steepening
     * Flat Pentacam keratometry reading ≥ 56.01 D
6. Presence of central or inferior steepening on the Pentacam map;
7. Have a maximum corneal curvature, as measured by Kmax of ≥ 47.00 D;
8. BSCVA (Best Spectacle Corrected Visual Acuity) of ≥ 1 letter and ≤ 80 letters on ETDRS (Early Treatment of Diabetic Retinopathy Study) chart;
9. Contact Lens Wearers Only: Removal of contact lenses is required for a 1 week period prior to the screening visit(s);
10. Contact Lens Wearers Only: Manifest refraction must be stable between two visits which occur at least 7 days apart. A stable refraction is one in which the manifest refraction spherical equivalent and the average K (Km) on the Pentacam taken at the first visit do not differ by more than 0.75 D from the respective measurements taken at the second exam.

Exclusion Criteria:

Patients must not meet any of he following criteria in order to be enrolled into the trial:

1. Contraindications, sensitivity or known allergy to the use of the test article(s) or their components;
2. If female, be pregnant, nursing or planning a pregnancy or have a positive urine pregnancy test prior to the randomization or treatment of either eye or during the course of the study;
3. Eyes classified as either normal, atypical normal, or keratoconus suspect on the severity grading scheme;
4. A history of previous corneal surgery or the insertion of Intacs in the eye to be treated;
5. A history of previous Limbal Relaxing Incision (LRI) procedure in the eye to be treated;
6. Corneal pachymetry that is < 375 microns prior to epithelial debridement at the thinnest point measured by Pentacam in the eye to be treated;
7. Eyes which are aphakic;
8. Eyes which are pseudophakic and do not have a UV blocking lens implanted;
9. Eyes that have the maximum corneal curvature (Kmax) outside of the central 5mm zone as measured by the Pentacam;
10. Previous ocular condition (other than refractive error) in the eye to be treated that may predispose the eye for future complications.

    For example:
    1. History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, corneal melt, corneal dystrophy, etc.);
    2. Clinically significant corneal scarring in the cross-linking treatment zone that is not related to keratoconus or, in the investigator's opinion, will interfere with the cross-linking procedure;
11. A history of delayed epithelial healing in the eye to be treated;
12. Patients with nystagmus or any other condition that would prevent a steady gaze during the treatment or other diagnostic tests;
13. Patients with a current condition that, in the investigator's opinion, would interfere with or prolong epithelial healing;
14. Taking Vitamin C (ascorbic acid) supplements within 1 week of the cross-linking treatment.
15. A history of previous corneal crosslinking treatment in the eye to be treated;
16. Have used an investigational drug or device within 30 days of the study or be concurrently enrolled in another investigational drug or device trial within 30 days of the study;
17. In addition, the Investigator may exclude or discontinue any subject for any sound medical reason.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Mean change in maximum corneal curvature (Kmax) between the VibeX active treatment group and placebo control group | baseline to 6 months

SECONDARY OUTCOMES:
Mean change in maximum corneal curvature (Kmax) between the VibeX active treatment group and placebo control group | baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vineeta Belanger, Study Director — Glaukos Corporation
Locations (10):
- United States (10):
  - UC Irvine Department of Ophthalmology, Irvine, California
  - Bascolm Palmer Eye Institute, Miami, Florida
  - Emory Eye Center, Atlanta, Georgia
  - Ophthalmic Consultants of Boston, Waltham, Massachusetts
  - Kugler Vision, Omaha, Nebraska
  - Pinceton Eye Goup, Princeton, New Jersey
  - Comprehensive Eye Care of Central Ohio, Westerville, Ohio
  - Medical University of South Carolina Storm Eye Institute, Magill Vision Center, Mt. Pleasant, South Carolina
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Hoopes Vision, Draper, Utah

IPD SHARING:
Plan to Share IPD: No